CLINICAL TRIAL: NCT05229783
Title: High Resolution Virtual Chromoendoscopy Versus Seattle Protocol for the Surveillance of Barrett's Esophagus: Impact on the Detection of High-grade Dysplasia and Adenocarcinoma Lesions
Brief Title: High Resolution Virtual Chromoendoscopy Versus Seattle Protocol for the Surveillance of Barrett's Esophagus
Acronym: CONVERSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: RC21_0411
Record Dates: First submitted 2021-12-07; First posted 2022-02-08 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Intervention Model Description: Each patient will be his (her) own control and have the two procedures :
  * Firsty : high-resolution endoscopy combined with virtual chromoendocopy (performed by endoscopist A)
  * Secondly: white light endoscopy with Seattle protocol (performed by endoscopist B)
Who Masked: Care Provider
Masking Description: The two endoscopists will be blinded to each other's findings when searching the lesions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic chromoendoscopy (Experimental): High-resolution endoscopy combined with virtual chromoendocopy to detect esophageal displasic lesions
  Interventions: Procedure: Electronic chromoendoscopy
- White light endoscopy with Seattle protocol (Active Comparator): White light endoscopy to detect esophageal displasic lesions, and then systemic quadrantic biopsies every 2 centimeters from the esogastric junction to the top of the Barett's esophagus (Seattle protocol)
  Interventions: Procedure: White light endoscopy with Seattle protocol

INTERVENTIONS:
Procedure: Electronic chromoendoscopy — Inspection of the Barrett's esophagus using the electronic chromoendoscopy modality of the endoscope for the detection of high-grade dysplasia and adenocarcinoma lesions.
  Arms: Electronic chromoendoscopy
Procedure: White light endoscopy with Seattle protocol — Inspection of the Barrett's esophagus using the white light modality of the endoscope for the detection of high-grade dysplasia and adenocarcinoma lesions, and then systemic quadrantic biopsies every 2 centimeters from the esogastric junction to the top of the Barett's esophagus (Seattle protocol)
  Arms: White light endoscopy with Seattle protocol

SUMMARY:
The investigators hypothesize that careful examination of Barrett's esophagus by high-resolution endoscopy combined with virtual chromoendoscopy could replace the Seattle protocol for Barrett's esophagus monitoring and detection of dysplasic lesions, and thus modify existing recommendations.

DETAILED DESCRIPTION:
Barrett's esophagus (BE) is a pre-neoplastic condition that predisposes to dysplasia and adenocarcinoma of the esophagus, a cancer with an increasing incidence and poor prognosis. However, when detected at an early stage, superficial lesions can be effectively treated by endoscopic resection. Although BE degeneration remains a rare event, the European Society for Gastrointestinal Endoscopy recommends that BE be followed according to its size. Follow-up consists of a digestive endoscopy with white light examination of the esophagus, targeted biopsies of any visible lesions and quadrantic biopsies every 2 centimeters from the esogastric junction to the top of the BE, at a frequency that depends on the presence of dysplasia and the size of the BE. However, physician adherence to this procedure, known as the Seattle Protocol, is low because : 1) it increases the time required for the endoscopist to examine the patient and therefore the duration of sedation, as well as the time needed to interpret the pathology, 2) the risk of sampling error is high because only a small portion of the esophageal mucosa can be biopsied and 3) this approach is costly because of the time spent on the Seattle protocol in the operating room and in the pathology department.

New optical tools such as high-resolution endoscopy combined with magnification and electronic chromoendoscopy can reveal subtle mucosal and microvascular changes in the BE, which could improve the detection of early neoplastic lesions. However, there is still insufficient evidence to recommend its use in routine BE surveillance.

The investigators hypothesize that careful examination of Barrett's Esophagus by high-resolution endoscopy combined with virtual chromoendoscopy could replace the Seattle protocol for BE monitoring and detection of dysplasic lesions, and thus modify existing recommendations.

In this study, each patient will be his(her) own control and have the two procedures :

* Firstly, an endoscopist called A will perform high-resolution endoscopy combined with virtual chromoendocopy and note on a scheme the biopsies/resection he would have done with this procedure.
* Secondly, another endoscopist called B will do the examination using white light modality of the endoscope and process as follows :

  1. He/she will describe all visible lesions with precise indications of their location on a virgin scheme;
  2. Then, he/she will be unblinded to endoscopist A findings, see the scheme of endoscopist A and perform biopsies/resection according to instructions of this scheme;
  3. He/she will perform the biopsies/resection he/she would have added (if any);
  4. Finally, he/she will perform the quadrantic biopsies according to Seattle Protocol.

Final histology results will serve as gold standard for the diagnosis of early esophageal adenocarcnoma or high grade displasia.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female with Age above ≥ years old;
* Female of childbearing potential must use appropriate method(s) of contraception during the clinical trial (i.e.: Intrauterine Device, pill, implant,sexual abstinence);
* Dysplastic Barrett's Esophagus preferably labelled "flat mucosal dysplasia";
* Patient requiring esophageal endoscopy as part of their regular monitoring;
* Affiliated to social security;
* Patient received Patient Information Form and accepted to participate to the study.

Exclusion Criteria:

* Previously treated Barrett's Esophagus;
* Known invasive esophageal adenocarcinoma;
* Contraindication to general anesthesia;
* Ongoing clopidogrel or anticoagulant therapy or coagulation disorder (platelet count < 50 000/mm3, Prothrombin time ratio <50%);
* Poor general health status precluding subsequent follow up of Barrett's Esophagus ;
* For female: pregnancy or breastfeeding;
* Adults under a legal protection regime (guardianship, trusteeship, "under judicial protection").
* Ongoing participation in another study requiring an intervention on Barrett's Esophagus during patient's participation in Converse study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Rate of both high grade dysplasia and esophageal adenocarcinoma lesions detected by electronic chromoendoscopy versus rate of such lesions detected by white light endoscopy plus systemic biopsies according to Seattle protocol. | Day 1

SECONDARY OUTCOMES:
Rate of both high grade dysplasia and esophageal adenocarcinoma lesions detected by electronic chromoendoscopy versus rate of such lesions detected by white light endoscopy. | Day 1
Rate of low grade displasia lesions detected by electronic chromoendoscopy versus rate of such lesions detected by white light endoscopy plus systemic biopsies according to Seattle protocol. | Day 1
Duration (in minutes) of each procedure: white light endoscopy, electronic chromoendoscopy, Seattle protocol. | Day 1
Rate of missed lesions (both high grade dysplasia and esophageal adenocarcinoma) diagnosed by an adjudication committee reviewing videos from the procedure. | Day 1
Rate of resected lesions (both high grade dysplasia and esophageal adenocarcinoma) that were detected by endoscopist performing electronic chromoendoscopy, but missed by endoscopist performing white light endoscopy and Seattle protocol. | Day 1
Number of adverse events | Day 30
Cost effectiveness of the detection of both early esophageal adenocarcinoma and high grade dysplasia with electronic chromoendoscopy versus cost effectiveness of Seattle protocol. | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Lucille QUENEHERVE, Doctor, Principal Investigator — CHU de Brest
Locations (15):
- France (15):
  - Amiens University Hospital, Amiens
  - Besançon University Hospital, Besançon
  - Bordeaux University Hospital, Bordeaux
  - Brest University Hospital, Brest
  - Private Bercy clinic, Charenton
  - Limoges University Hospital, Limoges
  - Lyon University Hospital, Lyon
  - Nancy University Hospital, Nancy
  - Nantes University Hospital, Nantes
  - Nice University Hospital, Nice
  - Public Assistance - Paris hospitals - Cochin hospital, Paris
  - Public Assistance- Paris Hospitals - Georges Pompidou European Hospital, Paris
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Sainte Barbe Clinic, Strasbourg

IPD SHARING:
Plan to Share IPD: No